CLINICAL TRIAL: NCT04111692
Title: A Prospective Observational Study of Foam Sclerotherapy for the Treatment of Symptomatic Kidney or Liver Cysts in Patients With Autosomal Dominant Polycystic Kidney and Liver Disease.
Brief Title: A Prospective Observational Study of Foam Sclerotherapy .
Status: Recruiting | Type: Observational
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Marie Hogan, Principal Investigator, Mayo Clinic
Other Study IDs: 17-006399
Record Dates: First submitted 2019-05-01; First posted 2019-10-01 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Autosomal Dominant Polycystic Kidney; Renal Cyst; Autosomal Dominant Polycystic Liver Disease; Hepatic Cyst
Keywords: hepatic cyst; Kidney Cyst; Autosomal Polycystic Liver Disease; Autosomal Polycystic Kidney Disease
MeSH Terms: conditions — Polycystic Kidney, Autosomal Dominant

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
An observational prospective study to determine the impact of foam sclerotherapy of large, dominant kidney/liver cysts on quality of life outcomes and kidney/liver cyst volumes at up to 12 months of follow-up in patients with autosomal dominant polycystic kidney disease (ADPKD) and autosomal dominant polycystic liver disease (ADPLD).

DETAILED DESCRIPTION:
Cyst burden is an important determinant of outcomes in both autosomal dominant polycystic kidney disease (ADPKD) (1, 2) and autosomal dominant polycystic liver disease (ADPLD) (3, 4). Furthermore, mass symptoms (from liver and kidney volume) greatly impact upon quality of life in patients with severe disease. Cyst volume increases exponentially with age and results in the development of end-stage renal disease and hypertension, compromised quality of life due to compressive symptoms, and predisposes patients to cyst complications such as infection, hemorrhage, rupture, and torsion. Existing percutaneous treatments for cyst burden in ADPKD and ADPLD include cyst aspiration with or without sclerotherapy. Although frequently effective in the short-term, recurrence rates and the need for repeat procedures are high after these procedures (5, 6). Extrarenal disease (primarily liver disease) is the most important aspect of disease burden to ADPKD patients (7), and there are few effective treatments.

Foam sclerotherapy (FS) with 3% Sodium Tetradecyl Sulfate (STS) a sclerosing agent. (Sotradecol®; Mylan, Galway, Ireland) is approved by the FDA for the management of varicose veins. While increasing cyst burden significantly compromises quality of life, the impact of FS on patient-reported outcomes has not been evaluated. In collaboration with the Center for Science of Healthcare delivery, we have developed a patient-reported outcome tool for polycystic liver disease capable of detecting symptom burden in individuals with polycystic liver disease that has been approved by the FDA as a patient-reported outcomes tool in research. Furthermore measurement of liver and kidney volumes can be performed in the Polycystic Kidney Disease Imaging Research Core that monitors organ volumes before and after interventions. At this time, patients are interested in procedures that will alleviate and palliate their mass symptoms but desire preliminary information on the procedural efficacy. We aim to report our experience with a new therapeutic advance - FS for the treatment of liver and kidney cysts at Mayo Clinic - and to determine the impact of this procedure on patient-reported quality of life measures and changes in organ volumes.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* Clinical diagnosis of ADPKD or ADPLD
* 1-3 large, non-exophytic liver or kidney cyst
* Compressive symptoms from dominant cyst

Exclusion Criteria:

* Age <18 years
* Absence of ADPKD or ADPLD
* Largest cyst <4cm in all 3 dimensions or largest cyst volume <400cc
* >3 large, non-exophytic liver or kidney cyst(s) ≥4cm in all 3 dimensions (cyst volume ≥400cc)
* Unwilling to comply with study follow-up protocol to 12 ± 1months post-FS
* Lacking capacity to provide informed consent to FS of liver or kidney cysts
* Pregnancy

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult subjects with ADPKD or ADPLD and large, symptomatic kidney or liver cysts followed in Nephrology or Hepatology clinics at Mayo Clinic, or de novo referrals to Mayo Clinic, Rochester, MN will be invited to participate.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2017-11-06 (Actual); Primary Completion 2027-11 (Estimated); Study Completion 2027-11 (Estimated)

PRIMARY OUTCOMES:
Change in Pain Inventory | Baseline, 1 month, 6 month, 12 month
  Measured using self assessed brief pain inventory (short form) questionnaire, using a scale of 0 is no pain and 10 is pain as bad as you can imagine
Change in Self Assessed Quality of life | Baseline, 1 month, 6 month, 12 month
  Measured using the linear analogue self assessed questionnaire, using a scale of 0 is as bad as it can be and 10 is as good as it can be
Change in health related quality of life | Baseline, 1 month, 6 month, 12 month
  Measured using the self assessed Medical Outcomes Study 36-Item Short-Form Health Survey (SF-36), using a scale that ranges from yes and no or all of the time to none of the time
Change in Polycystic Liver Disease Quality of Life | Baseline, 1 month, 6 month, 12 month
  Measured using the self assessed Polycystic Liver Disease Questionnaire, using a scale that ranges from never/not at all to always/a lot

CONTACTS AND LOCATIONS:
Overall Officials: Marie Hogan, MD, PhD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials